CLINICAL TRIAL: NCT05723666
Title: The Effect of Virtual Reality Glasses on Fear of Birth, Delivery Time and Non-Stress Test Results in Pregnancy in the Process of Labor: A Randomized Controlled Single-Blind Study
Brief Title: The Effect of Virtual Reality Glasses on Fear of Birth, Delivery Time and Non-Stress Test Results in Pregnancy in the Process of Labor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Mine ORUC, Lecturer, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Mine ORUÇ; Kamile KABUKCUOĞLU (Other: Akdeniz University)
Record Dates: First submitted 2022-01-21; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Virtual Reality
Keywords: virtual reality; fear of childbirth; non-stress test; time of delivery

STUDY DESIGN:
Intervention Model Description: There are two Groups with parallel properties. The first group is the experimental group using virtual reality glasses.
  The second group is the control group without intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group watching video with virtual reality glasses (Experimental): A nature video will be watched with virtual reality glasses.
  Interventions: Other: Group watching virtual reality glasses
- Group not watching video with virtual reality glasses (No Intervention): Virtual reality glasses will not be watched. An intervention will not be applied.

INTERVENTIONS:
Other: Group watching virtual reality glasses — A nature video will be watched with virtual reality glasses.
  Arms: Group watching video with virtual reality glasses

SUMMARY:
From the gestation period, labor affects the mother due to both physical and emotional changes. Mothers experience new emotions and experiences since their admission to the delivery room. With the progression of the mother's physiological changes and labor in the delivery room, new situations arise. Although the birth process is a complex process, it can vary from person to person. In the delivery room, many preparations and applications are made for labor. A positive pregnancy and childbirth will affect both the motherhood process and later life periods. Every day, new applications are added to the applications made for the mother to leave the labor satisfied. Virtual reality (VR) glasses application has features such as relaxation, distraction, reducing focus on pain, painful and stressful applications. When the literature is examined, SG glasses are generally focused on pain in the field of women's health. In this study, it is aimed to evaluate the effect of watching videos with SG glasses on the fear of childbirth, NST results and delivery time by using the distraction feature of the mother in the delivery room. The study included mothers who came to Antalya Training and Research Hospital delivery room for vaginal delivery, aged 18-35, had no hearing and vision problems, had an uneventful pregnancy, and had no chronic disease in the fetus or mother. A total of 128 mothers with 64 experimental (32 primiparous, 32 multiparous), 64 control groups (32 primiparous, 32 multipara) and a total of 128 mothers will be included in the study by power analysis. For the randomization of this study, which was planned as a randomized controlled trial, "simple randomization method" stratified sampling, which was admitted to the delivery room and met the inclusion criteria, was used. In the study, mothers in the experimental group will be shown a nature video with SG glasses during the NST procedure. No intervention other than routine delivery room care will be applied to the control group. At the end of the study, it is expected that the level of fear of birth will decrease, the NST will be reactive, and the duration of labor will decrease with the relief of the mothers' SG glasses.

DETAILED DESCRIPTION:
The birth of a baby is expressed as a unique life experience for every mother. From the pregnancy period, labor affects the mother to a great extent due to both physical and emotional changes. Mothers experience new emotions and experiences since their admission to the delivery room. Birth is a situation where fear, sadness, pain, happiness and joy are experienced together. For this reason, the practices made since the admission of women to the delivery room include an unforgettable experience in women's life.

Labor takes place in a total of four stages, including the onset and completion of effacement and dilatations, the tightening of contractions, the birth of the baby, the birth of the placenta and membranes, and the first four hours afterward. Although the duration of delivery may vary in multiparous and primiparous cases, it should not exceed 24 hours. It has been reported that pregnant women admitted to the delivery room before the active phase stay in the delivery room more, spend labor alone, face more negative situations, and have more stress due to monitoring and analgesia.

Fetal monitoring, induction application, enema, cervical examination, use of analgesia to reduce labor pain for monitoring maternal and fetal health during labor, Applications such as bladder catheter, episiotomy, dose and duration of epidural anesthesia are performed and these applications directly affect the duration of delivery and the length of stay of the mother in the delivery room. Despite all these practices, it is not yet known what the most effective and successful method for initiating and accelerating labor is. In addition to the pharmacological and mechanical methods applied, non-pharmacological and supportive care practices in labor, which are more preferred by women, are also being developed.

In recent years, the idea that childbirth is a natural process that is disrupted by medical interventions has become increasingly common. If the needs of the pregnant woman are known and respected during labor, it is aimed to reduce the need for non-medical supportive care, which facilitates the pregnant woman to use coping methods more, and aims to reduce her anxiety, discomfort, loneliness and fatigue, and to reduce excessive and unnecessary interventions. The use of applications for non-pharmacological care in the labor process is increasing day by day. Acupressure, acupuncture, music therapy, massage treatments, breathing techniques, yoga, hypnosis. Methods such as focusing, distraction, daydreaming, hydrotherapy can be used. Non-pharmacological methods do not prolong the delivery period and attract attention as they have no side effects, no allergy risk, are economical, reliable and easy to use. There is a need for further development of these methods, which are found by trial and error in different countries.

From the mother's admission to the delivery room, many preparations and practices are made for labor. Non-invasive non-stress testing (NST) is frequently used in the evaluation of the well-being of the mother and the baby in the delivery room. The nonstress test is a test used to monitor the heartbeat of the fetus, and to determine the relationship between fetal movements and uterine contractions, if any. The NST is evaluated for at least 20 minutes while the expectant mother is lying on her back or on her left side. A reactive NST is expected to have at least 2 accelerations within 20 minutes and short-term variability to be moderate. NST without at least 2 accelerations for 20 minutes, up to 40 minutes If it still fails, it is considered as non-reactive NST. NST is one of the most important methods used in pregnancy follow-ups to show fetal well-being. The most important disadvantage is the need for further extension of the test period and repetition due to reasons such as long application time and non-reactive NST. The NST can be affected by the mother's intake of sufficient fluid, the mother's hunger or satiety, drug or smoking status, excitement, fear and stress level, and the noise level of the environment. Many non-pharmacological methods are tried to improve maternal and fetal outcomes in NST. It has been reported that music, stress and anxiety during the NST procedure, relaxing hypnotherapy, and distraction methods reduce anxiety in pregnant women and lead to an increase in the number of fetal movements and accelerations.

Pain due to contractions during labor, experiences related to the moment of birth, birth stories heard from others, uncertainty, mother's stress state, routine care given in the delivery room cause fear and stress. Practices in the delivery room, loneliness due to the length of stay and uncontrollable psychological support may cause fear of childbirth in pregnant women. Fear of childbirth; It is an anxiety that starts before pregnancy and includes the fear of birth and death. This situation, which may differ in every woman, cause negative consequences in women, and intensify gradually, is defined as "Tokophobia". Other important reasons that trigger the fear of childbirth; Problematic birth experiences such as risky pregnancy history, listening to or watching fearful experiences of others, difficult labor with vacuum or forceps intervention, history of anomaly or stillbirth, history of excessive blood loss during delivery, emergency cesarean section decision, emergencies during delivery is the mother's inability to receive adequate social support during pregnancy and delivery.

Prevalence of fear of childbirth in pregnant women; sociodemographic, obstetric and cultural differences. Not knowing the methods of coping with the fear of childbirth further complicates the situation. It is known that the care given in the delivery room shortens the duration of labor, reduces the fear of childbirth, is exposed to less pharmacological support and obstetric intervention, decreases the risk of perinatal complications, episiotomy application, oxytocin use and cesarean section rates. As non-pharmacological methods to reduce fear of childbirth, breathing exercises, hydrotherapy, meditation, breathing exercises, daily walks, hypnotic birth, yoga, social support and birth information training given in pregnant schools were found to be effective in reducing fear of birth .

Although most women describe childbirth as a powerful and positive experience, some women may feel helpless, detached from life and abandoned during childbirth. Stress, anxiety, fear, labor pain, fear of the unknown regarding childbirth, distrust of caregivers increase the secretion of catecholamines, cortisone and epinephrine. For this reason, the duration of delivery, non-stress test results and fear of childbirth are negatively affected. In recent years, simple and easy non-pharmacological methods to manage these conditions and reduce negative effects have come to the fore. Distraction methods are focused on the basis of the non-pharmacological methods applied.

Distraction is focusing one's attention from the current situation to another situation. It is used in many ways for distraction. There is information that listening to music, watching videos, exercising, reading a book, breathing techniques or handicraft activities attract attention at a substantial level. The person can distance himself from situations such as fear, stress and anxiety, which he feels with distraction methods. Regardless of the method used, distraction helps to relax and get away from stress.

World Health Organization, technology in health services; It is defined as the application of organized knowledge and capabilities developed through systems, vaccines, drugs, devices developed to improve quality of life and solve health problems. It is reported that these devices have been developed to increase the quality of care, to correct or change body functions, apart from the purposes such as the prevention, diagnosis and treatment of diseases. In recent years, new technologies have been used in the care applied in nursing services. Virtual reality (Virtual Reality/VR) has many application areas related to care and treatment in the health sector. VR technology is used as a tool to support surgery, health care services, rehabilitation of patients and exercise, education of patients, healthcare workers and clinical students, and preventive and caregiver health services in clinical applications.

Virtual reality is defined as "a technology that gives the feeling that three-dimensional pictures and animations created in the computer environment are in a real environment in people's minds with technological tools and enables them to interact with these objects in the environment". It usually allows the person to interact in this new world, by using technology to create a dimension that the person experiences as reality in the virtual environment. The purpose of VR is to make the user believe that they are in a computer-generated environment as much as possible. VR simulators are technically advanced and available in a variety of sizes and shapes. VR provides a three-dimensional environment, including a head-mounted device, 3D-capable glasses, headsets, and/or other similar sensors. Thanks to its audio and visual settings, it is possible to interact with a simulated, lifelike or fantastic environment.

Virtual reality glasses (Visual Reality-VR) are used as a tool to support preventive health services in clinical applications. VR, which is among the technological products, can be used in non-pharmacological methods as well as pharmacological methods. Although there are discussions about the harms and benefits of non-pharmacological use, there are many studies in the literature showing that it is effective. The effect is directly proportional to the level of the patient in the virtual environment. Patient interaction is a uniquely effective method of distraction (compared to video or audio stimulation) as it is multidimensional, immersive, and interactive. In general, VR has been described as an effective tool for distraction in medical procedures.

One of the recent uses of virtual reality is women's health. Studies in this area have found that virtual reality is an effective non-pharmacological method to reduce pain and anxiety during labor. It is stated that daydreaming or music during labor has an effect on distraction and relaxation. However, because sometimes dreaming and dreaming can be difficult for women, watching videos with virtual reality glasses is a good alternative.

Life is a continuous process, each phase of which affects the next. Childbirth and motherhood are considered the most important stages of a woman's life. A positive pregnancy and childbirth will affect both the motherhood process and later life periods. Every day, new applications are added to the applications made for the mother to leave the labor satisfied. Virtual glasses application has features such as relaxation, distraction, reducing focus on pain and painful applications. In this study, it is aimed to evaluate the effect of fear of childbirth, NST results, and duration of delivery by watching the video with virtual reality glasses in the delivery room, distracting the mother's attention and providing relaxation.

ELIGIBILITY:
Inclusion Criteria:

* Verbal communication,
* Between the ages of 20 and 35,

  ·-No limitation of hearing and vision,
* Gestational week between 35-42,
* Vaginal delivery planned,
* Do not have any risk factors (premature rupture of membranes, preeclampsia, gestational diabetes, etc.) during pregnancy,
* No defined cardiovascular disease, anomaly, IUGR (intrauterine growth retardation) in the fetus,

Exclusion Criteria:

* Diagnosed with risky pregnancy,
* Having obstetric complications,
* Have a previous negative birth history,
* Having a psychiatric diagnosis,
* Have a systemic disease,
* Those who watch the video for less than 20 minutes,
* Those who went to the cesarean operation,
* Those with positive or symptomatic COVID-19 PCR test

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women
Enrollment: 128 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
physiological parameter | 48 hour
  reactive NST,
Wijma Delivery Expectancy/Experience Questionnaire (W-DEQ) Version A and B | 48 hour
  low fear of childbirth
physiological parameter | 2 hour
  positive effects on labor time

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No